CLINICAL TRIAL: NCT01968434
Title: Randomized, Single Blind, Multicenter Study to Evaluate the Efficacy and Tolerability of Syr. Grintuss Pediatric and Syr. Mucolit in Cough Due to Upper Respiratory Tract Infection in Children
Brief Title: Comparison of Efficacy and Tolerability of Two Cough Syrups in Cough Due to Cold in Children.
Acronym: URTI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clalit Health Services (Other)
Collaborators: Aboca Spa Societa' Agricola (Industry)
Responsible Party: Principal Investigator, Avner Herman Cohen, MD. Head Dep. Pediatric Ambulatory Clinic -Petah-Tikva, Israel, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COM-13-00
Record Dates: First submitted 2013-10-17; First posted 2013-10-24 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Cough; Upper Respiratory Tract Infection
Keywords: cough; common cold; antitussive agents; mucosal protection; medical device
MeSH Terms: conditions — Cough; Respiratory Tract Infections; Common Cold

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- protective cough syrup (Experimental): syrup containing honey, plantago lanceolata, grindelia robusta, helichrysum italicum ina syrup form. The cough syrup is a CE marked medical device acting in a non pharmacological way to reduce cough.
  Dosage: 20 ml divided in three doses per day for the duration of the study (4 nights, 3 days)
  Interventions: Device: protective cough syrup
- carbocisteine cough syrup (Active Comparator): Dosage 20-25 mg/kg/day three times a day (3 days/4 nights)
  Interventions: Drug: carbocisteine cough syrup

INTERVENTIONS:
Device: protective cough syrup — The mucoadhesive and radical scavenging properties of the components create a protective film on the pharynx which protects irritated mucosa from cough generating stimuli such as post nasal drip, irritating elements, dehydration.
  Other Names: Grintuss
  Arms: protective cough syrup
Drug: carbocisteine cough syrup — Mucolytic
  Other Names: Mucolit; Lisomucil
  Arms: carbocisteine cough syrup

SUMMARY:
The purpose of this study is to determine if there is comparable efficacy between carbocisteine and a protective cough syrup from natural ingredients in children's cough due to upper respiratory tract infections (URTI) such as the common cold. The hypothesis is that protecting the throat is very useful in decreasing cough severity, both day and night, without needing to subdue such an important reflex as cough, and without only acting on mucous fluidification, especially in children where sedation and excessive fluidification is dangerous. The research hypothesis is that the protective (Grintuss) Syrup relieves cough (frequency, intensity, degree of disturbance due to nocturnal cough, and improves the quality of sleep of the child) as much as or more than the carbocysteine syrup usually used to treat children (Syr Mucolit).

DETAILED DESCRIPTION:
Cough is a life saving reflex, therefore it is important, especially in pediatrics, to calm cough spells without sedating the reflex. Mucolytic agents have been shown to be helpful but side effects have been reported and use has been prohibited under 2 years of age. Therefore, a completely safe and effective cough remedy has not been officially reported yet in a randomised trial. Looking into other mechanisms for cough management such as protection of irritated pharynx mucosa from post nasal drip or other irritating substances is theoretically sound and shows practical interesting results.

A parallel comparison of efficacy and tolerability between such protective mechanism (acting through a barrier and radical scavenging action) due to natural substances (honey, plantago lanceolata, grindelia robusta and helichrysum italicum) and a mucolytic substance has not been done so far, in young children, especially in a time frame of 4 days. The intent of this study is to use the protective syrup versus carbocysteine in children with moderate to severe night and daily cough, measured with a validated parent questionnaire. The invasiveness of cough is followed immediately after one night administration of the study products and daily for four days.

A similar effectiveness of the protective cough syrup as compared to carbocisteine is considered very interesting due to the mechanism of the remedy.

ELIGIBILITY:
Inclusion Criteria:

* cough attributed to URTI such as the common cold
* 2-5 years of age
* moderate to severe day cough according to questionnaire (score at least 3 on all 3 questions relating to day cough) considering the day prior to enrollment.
* moderate to severe night cough score according to questionnaire (score at least 3 of 2 of the three questions relating to the evaluation of nocturnal cough (frequency of nocturnal cough, impact of the sleep of the child and impact on the sleep of the parent)
* signature of informed consent

Exclusion Criteria:

* Children with the diagnosis of diseases of the lower respiratory tract: inflammation of the larynx, trachea, bronchi, pneumonia, asthma, sinusitis, allergic rhinitis, as well as heart disease.
* Children who received cough medicines or drugs containing antihistamines the day prior to study entry.
* Known hypersensitivity to honey or any other component of the experimental product such as Grindelia, Helichrysum, essential oils natural flavourings of Lemon, Sweet Orange, Myrtle; Lemon natural flavouring
* Children who received any steroid preparation (spray nozzle , or syrup , or other similar the day before study entry )
* Known sensitivity to carbocysteine specifically to the comparator Mucolit
* gastric ulcer

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Avner Cohen, Professor, Principal Investigator — Clalit Health Services
Locations (4):
- Israel (4):
  - Pediatric Ambulatory Clinic Bat-Yam, Bat Yam
  - Pediatric Ambulatory Clinic Kfar-Saba, Kfar Saba
  - Pediatric Community Ambulatory Clinic - Petach-Tikva, Petah Tikva
  - Pediatric Ambulatory Clinic Ramat Aviv Gimel, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Middleton KR, Hing E. National Hospital Ambulatory Medical Care Survey: 2004 outpatient department summary. Adv Data. 2006 Jun 23;(373):1-27. PMID 16841784
- [Background] Paul IM, Yoder KE, Crowell KR, Shaffer ML, McMillan HS, Carlson LC, Dilworth DA, Berlin CM Jr. Effect of dextromethorphan, diphenhydramine, and placebo on nocturnal cough and sleep quality for coughing children and their parents. Pediatrics. 2004 Jul;114(1):e85-90. doi: 10.1542/peds.114.1.e85. PMID 15231978
- [Background] Paul IM, Beiler J, McMonagle A, Shaffer ML, Duda L, Berlin CM Jr. Effect of honey, dextromethorphan, and no treatment on nocturnal cough and sleep quality for coughing children and their parents. Arch Pediatr Adolesc Med. 2007 Dec;161(12):1140-6. doi: 10.1001/archpedi.161.12.1140. PMID 18056558
- [Background] Department of child and adolescent health. Cough and cold remedies for the treatment of acute respiratory infections in young children. Geneva, Switzerland: World Health Organization: 2001.
- [Background] Allen KL, Molan PC, Reid GM. A survey of the antibacterial activity of some New Zealand honeys. J Pharm Pharmacol. 1991 Dec;43(12):817-22. doi: 10.1111/j.2042-7158.1991.tb03186.x. PMID 1687577
- [Background] Schramm DD, Karim M, Schrader HR, Holt RR, Cardetti M, Keen CL. Honey with high levels of antioxidants can provide protection to healthy human subjects. J Agric Food Chem. 2003 Mar 12;51(6):1732-5. doi: 10.1021/jf025928k. PMID 12617614
- [Background] Cohen HA, Rozen J, Kristal H, Laks Y, Berkovitch M, Uziel Y, Kozer E, Pomeranz A, Efrat H. Effect of honey on nocturnal cough and sleep quality: a double-blind, randomized, placebo-controlled study. Pediatrics. 2012 Sep;130(3):465-71. doi: 10.1542/peds.2011-3075. Epub 2012 Aug 6. PMID 22869830
- [Background] Bogdanov S, Jurendic T, Sieber R, Gallmann P. Honey for nutrition and health: a review. J Am Coll Nutr. 2008 Dec;27(6):677-89. doi: 10.1080/07315724.2008.10719745. PMID 19155427
- [Background] Rimsza ME, Newberry S. Unexpected infant deaths associated with use of cough and cold medications. Pediatrics. 2008 Aug;122(2):e318-22. doi: 10.1542/peds.2007-3813. PMID 18676517
- [Background] Kraft K. Efficacy of fluid in Plantago lanceolata extract (PLFE) in acute respiratory disease. Phytomedicine, Supplement 1, 1996
- [Background] Wegener T, Kraft K. [Plantain (Plantago lanceolata L.): anti-inflammatory action in upper respiratory tract infections]. Wien Med Wochenschr. 1999;149(8-10):211-6. German. PMID 10483683

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting took place within the Clalit health service community day hospitals. Community day hospitals are places where parents go for usual illnesses and treat most community ailments.
Pre-assignment Details: Access for eligibility= 195 Excluded =45 (refused to participate n= 24, not meeting inclusion criteria n=21)
Groups:
- Protective Cough Syrup: syrup containing honey, plantago lanceolata, grindelia robusta, helichrysum italicum ina syrup form. The cough syrup is a CE marked medical device acting in a non pharmacological way to reduce cough.
  Dosage: 6,5 ml three times a day for the duration of the study (4 nights, 3 days)
  protective cough syrup: The mucoadhesive and radical scavenging properties of the components create a protective film on the pharynx which protects irritated mucosa from cough generating stimuli such as post nasal drip, irritating elements, dehydration.
  Access for eligibility= 195 Excluded =45 (refused to participate n= 24, not meeting inclusion criteria n=21) Enrolled: 150 completed pre-treatment questionnaire and randomized into groups Allocated protective syrup n = 78 received intervention n= 78 Lost to follow up n=3 Discontinued intervention n=0 Analyzed n=75 Excluded from analysis n=0
- Carbocisteine Cough Syrup: Dosage 20-25 mg/kg/day three times a day (3 days/4 nights)
  carbocisteine cough syrup: Mucolytic
  Access for eligibility= 195 Excluded =45 (refused to participate n= 24, not meeting inclusion criteria n=21) Enrolled: 150 completed pre-treatment questionnaire and randomized into groups Allocated carbocisteine syrup n = 72 received intervention n= 72 Lost to follow up n=6 Discontinued intervention n=0 Analyzed n=66 Excluded from analysis n=0
Period: Overall Study
Arm/Group | Protective Cough Syrup | Carbocisteine Cough Syrup
Started | 78 | 72
Completed | 75 | 66
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Population: Enrolled patients had a minimum cough intensity both day and night, according to questionnaire, had not received any cough medicine the day before enrollment and fulfilled all inclusion criteria.
Groups:
- Protective Cough Syrup: syrup containing honey, plantago lanceolata, grindelia robusta, helichrysum italicum in a syrup form. The cough syrup is a CE marked medical device acting in a non pharmacological way to reduce cough.
  Dosage: 6.5 ml three times a day for the duration of the study (4 nights, 3 days)
  protective cough syrup: The mucoadhesive and radical scavenging properties of the components create a protective film on the pharynx which protects irritated mucosa from cough generating stimuli such as post nasal drip, irritating elements, dehydration.
  Enrolled: 150 completed pre-treatment questionnaire and randomized into groups Allocated protective syrup n = 78 received intervention n= 78 Lost to follow up n=3 Discontinued intervention n=0 Analyzed n=75 Excluded from analysis n=0
- Carbocisteine Cough Syrup: Dosage 20-25 mg/kg/day three times a day (3 days/4 nights)
  carbocisteine cough syrup: Mucolytic
  Enrolled: 150 completed pre-treatment questionnaire and randomized into groups Allocated carbocisteine syrup n = 72 received intervention n= 72 Lost to follow up n=6 Discontinued intervention n=0 Analyzed n=66 Excluded from analysis n=0
- Total: Total of all reporting groups
Arm/Group | Protective Cough Syrup | Carbocisteine Cough Syrup | Total
Number analyzed (Participants) | 78 | 72 | 150
Age, Continuous [Mean (Standard Deviation); unit: months] | 42.49 (12.96) | 43.17 (14.57) | 42.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 37 | 34 | 71
Region of Enrollment [Number; unit: participants]
  Israel | 78 | 72 | 150
Participants coughing since ≥ 3 days at time of enrollment [Number; unit: participants] | 47 | 46 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change in Night Cough Score on First Night of Treatment (From N0 to N1)
Description: Night cough is most bothersome to the child and family. Cough was measured with a validated questionnaire which asks parents to rate 5 aspects of night cough: frequency, severity, bothersomeness, child sleep and parent sleep according to a 7 point Likert scale, from 0 (not at all) to 6 (extremely). Lower scores indicate a better condition. The morning after the first night of treatment (N1) the parents rated the passed night by scoring from 0-6 each of the 5 aspects of night cough. The sum of scores for all 5 aspects gives the combined night cough score. This score, ranging between 0-30, was subtracted from the sum of all aspects, also ranging between 0-30, form the basal night cough score of the night before enrollment (N0). This change is recorded as "change in combined night cough score" and it refers to the change from N0 to N1. Negative values of the change indicate an improvement in the condition of the patient.
Time Frame: 1 night from before enrollment (N0) to first night after treatment (N1)
Population: the population analyzed are the children who completed the protocol and submitted the complete questionnaire for night and day cough. 78 patients were enrolled in the protective syrup Group and 72 in the carbocysteine Group. 3 patients in the protective syrup group and 6 in the carbocysteine group never began the study.
Measure: Mean (Standard Error); unit: change in combined night cough score
Groups:
- Protective Cough Syrup: syrup containing honey, plantago lanceolata, grindelia robusta, helichrysum italicum ina syrup form. The cough syrup is a CE marked medical device acting in a non pharmacological way to reduce cough.
  Dosage: 20 ml divided in three doses per day for the duration of the study (4 nights, 3 days)
  protective cough syrup: The mucoadhesive and radical scavenging properties of the components create a protective film on the pharynx which protects irritated mucosa from cough generating stimuli such as post nasal drip, irritating elements, dehydration.
Arm/Group | Protective Cough Syrup | Carbocisteine Cough Syrup
Number analyzed (Participants) | 75 | 66
change in combined night cough score | -5.16 (0.85) | -1.77 (0.67)
Statistical Analysis 1: Comparison: Protective Cough Syrup vs Carbocisteine Cough Syrup; The sample size was calculated to detect a 0.75 point difference between any two treatment groups with a 90% power and p<0.05. Such sample size was 60 subject which was elevated ot 75 subjects per group to account for drop outs. For comparison of cough evaluation before and after treatment a paired Student t test was used; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Change in Night Cough Score at End of Study (From N0 to N4)
Description: A validated cough questionnaire measuring 5 aspects of night cough (frequency, severity, bothersomeness, child sleep and parents' sleep) on a 7 point Likert scale was used each morning to rate the passed night. The scale rates each parameter from 0 (not at all) to 6 (extremely). Every night of the trial is rated. The morning after the last night of the study (N4) the parents rated the passed night by scoring from 0-6 each of the 5 aspects of night cough. The summed score for all aspects gives the combined night cough score. This score, ranging between 0-30, was subtracted from the sum of all aspects, also ranging between 0-30, form the basal night cough score of the night before enrollment (N0). This change is recorded as "change in combined night cough score" and it refers to the change from N0 to N4. Negative values of the change indicate an improvement in the condition of the patient.
Time Frame: 4 nights (onset of trial Night 1 to Night 4) and 3 days
Population: 78 patients were enrolled in the protective syrup Group and 72 in the carbocysteine Group. 3 patients in the protective syrup group and 6 in the carbocysteine group never began the study. 7 patients from the protective syrup group and twelve 12 patients from the carbocysteine group did not answer the questions for the last night.
Measure: Mean (Standard Error); unit: change in combined night cough score
Arm/Group | Protective Cough Syrup | Carbocisteine Cough Syrup
Number analyzed (Participants) | 71 | 60
change in combined night cough score | -13.92 (0.92) | -9.48 (1.08)
Statistical Analysis 1: Comparison: Protective Cough Syrup vs Carbocisteine Cough Syrup; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

3. Secondary Outcome: Change in Day Cough Score at End of Study (From D0 to D4)
Description: A validated cough questionnaire measuring 3 aspects of daytime cough (frequency, severity, bothersomeness) on a 7 point Likert scale was used each evening to rate the passed day, as regards these aspects. The scale rates each parameter from 0 (not at all) to 6 (extremely). Every day of the trial is rated. The last evening of the study (D4) the parents rated the passed day by scoring from 0-6 each of the 3 aspects of day cough. The summed score for all aspects gives the combined day cough score. This score, ranging between 0-18, was subtracted from the sum of all aspects, also ranging between 0-18, form the basal day cough score of the day before enrollment (D0). This change is recorded as "change in combined day cough score" and it refers to the change from D0 to D4. Negative values of the change indicate an improvement in the condition of the patient.
Time Frame: 4 nights (onset of trial Night 1 to Night 4) and 3 days
Population: 78 patients were enrolled in the protective syrup Group and 72 in the carbocysteine Group. 3 patients in the protective syrup group and 6 in the carbocysteine group never began the study. 6 patients from the protective syrup group and twelve 11 patients from the carbocysteine group did not answer the questions for the last day.
Measure: Mean (Standard Error); unit: change in combined day cough score
Arm/Group | Protective Cough Syrup | Carbocisteine Cough Syrup
Number analyzed (Participants) | 72 | 61
change in combined day cough score | -6.17 (0.43) | -4.54 (0.6)
Statistical Analysis 1: Comparison: Protective Cough Syrup vs Carbocisteine Cough Syrup; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during study period, from first enrollment to last collected data, which was a period of 5 months. Due to the nature of ailment and of treatment it was envisaged that any adverse event would be evident within study period.
Description: Adverse events were systematically collected by the CRF questionnaire.
Groups:
- Protective Cough Syrup: syrup containing honey, plantago lanceolata, grindelia robusta, helichrysum italicum ina syrup form. The cough syrup is a CE marked medical device acting in a non pharmacological way to reduce cough.
  Dosage: 6,5 ml three times a day for the duration of the study (4 nights, 3 days)
  protective cough syrup: The mucoadhesive and radical scavenging properties of the components create a protective film on the pharynx which protects irritated mucosa from cough generating stimuli such as post nasal drip, irritating elements, dehydration.
Arm/Group | Protective Cough Syrup | Carbocisteine Cough Syrup
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/66
Other Adverse Events (participants affected / at risk) | 6/75 | 9/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protective Cough Syrup (N=75) | Carbocisteine Cough Syrup (N=66)
nausea (Gastrointestinal disorders) | 5 (5) | 6 (6)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
drowsiness (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No